CLINICAL TRIAL: NCT02034968
Title: Nimotuzumab Plus Nab-paclitaxel and Cisplatin in Treating Patients With Advanced Esophageal Carcinoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No recruitment
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Qiong Zhao, Chief of Department of Thoracic Oncology, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZYTOP1406
Record Dates: First submitted 2014-01-10; First posted 2014-01-14 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Stage IV Esophageal Squamous Cell Carcinoma
Keywords: Nimotuzumab; Nab-Paclitaxel; Carcinoma of Esophagus
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma; Esophageal Neoplasms | interventions — nimotuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nimotuzumab & nab-paclitaxel & cisplatin (Experimental): Nimotuzumab: 200mg,IV once a week during chemotherapy.
  Nab-paclitaxel: 125mg/m2,(IV over 30 min) (days 1 and 8) on 21 day cycle
  Cisplatin: 75mg/m2,IV on 21 day cycle
  Interventions: Drug: Nimotuzumab

INTERVENTIONS:
Drug: Nimotuzumab — Nimotuzumab: 200mg,IV once a week during chemotherapy.
  Other Names: Anti epidermal growth factor receptor antibody h-R3

SUMMARY:
There have been reports suggesting that anti-epidermal growth factor antibody nimotuzumab is advantageous for advanced esophageal cancer patients in combination with chemotherapy or radiotherapy.And,albumin-bound paclitaxel was characterized with high tolerated doses with greater efficacy,and with greater concentration in tumor tissue compared with normal tissues.So,The objective of this single-arm phase II trial was to evaluate the benefit of nimotuzumab plus nab-paclitaxel and cisplatin in patients with advanced esophageal carcinoma.

DETAILED DESCRIPTION:
In the past decade, clinical trials have evaluated the role of chemotherapy, radiation, or both, for patients with advanced esophageal carcinoma, but have all failed to demonstrate a consistent survival benefit. In Eastern countries, Chemotherapy became one of the treatment strategies for advanced esophageal cancer. In an effort to improve the efficacy of systemic chemotherapy, the investigators conducted a prospective study to evaluate the regimen of Nimotuzumab plus Nab-paclitaxel/cisplatin for patients with advanced esophageal squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Patient who was confirmed stage IV esophageal carcinoma by pathologic histology or cytology.
* Males or females aged ≥18 years, < 75 years.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Life expectancy ≥12 weeks.
* Adequate bone marrow, renal, and liver function are required.
* Able to comply with the required protocol and follow-up procedures, and able to receive oral medications.

Exclusion Criteria:

* Any unstable systemic disease (including active infection, uncontrolled hypertension, unstable angina, congestive heart failure, myocardial infarction within the previous year, serious cardiac arrhythmia requiring medication, hepatic, renal, or metabolic disease).
* Allergy to anti-EGFR antibody.
* Female subjects should not be pregnant or breast-feeding.
* Adequate hematological function: Absolute neutrophil count (ANC) ≥1.5 x 109/L, and Platelet count ≥100 x 109/L. Adequate renal function: Serum creatinine ≤ 1.5 x ULN, or ≥ 50 ml/min. Adequate liver function: total bilirubin < 1.5 x upper limit of normal (ULN) and alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5 x ULN in the absence of liver metastases, or < 5 x ULN in case of liver metastases.
* Patient assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-02; Primary Completion 2016-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival(PFS) | 12 months

SECONDARY OUTCOMES:
Objective Response Rate | From date of treatment until the date of progression, assessed up to 2 months

OTHER OUTCOMES:
Overall survival (OS) | 12 months
Adverse events | During the chemotherapy,an expected average of 3 weeks
  Adverse events were classified according to U.S. National Cancer Institute common toxicity criteria, version 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Qiong Zhao, MD, Principal Investigator — The First Affiliated Hospital, Zhejiang University
Locations (1):
- The first affiliated hospital, Zhejiang University, Hangzhou, Zhejiang, China